CLINICAL TRIAL: NCT05943171
Title: A Randomized Controlled Trial of A Digital, Self-Guided, Avatar Assisted- Cognitive Behavioral Therapy Platform to Treat Addiction: RITch®CBT vs. Treatment As Usual
Brief Title: A Randomized Controlled Trial of Digital CBT to Treat Addiction: Digital RITch®CBT vs. Standard CBT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Caroline Easton, Academic Division Chief of Addiction Psychiatry, Professor of Psychiatry, Director of Digital Therapeautics, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00010815; 7UG3DA057042-03 (NIH)
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorders; Alcohol Use Disorder; Stimulant-Related Disorder
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism

STUDY DESIGN:
Intervention Model Description: Randomized to either Digital Avatar Assisted CBT or Human Administered CBT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Digital RITch®CBT (Experimental): (Digital RITch®CBT) is a Digital Avatar Assisted Interactive CBT Treatment
  Interventions: Device: Cognitive Behavioral Therapy
- Human Administered CBT (Active Comparator): Standard CBT is a human administered CBT Treatment
  Interventions: Behavioral: Standard CBT

INTERVENTIONS:
Device: Cognitive Behavioral Therapy — Digital treatment that deploys CBT.
  Other Names: Device (Digital RITch®CBT)
  Arms: Digital RITch®CBT
Behavioral: Standard CBT — Human Administered Manualized CBT
  Arms: Human Administered CBT

SUMMARY:
Substance Use Disorders continue to increase across the United States with significant adverse effects resulting in more than $700 billion annually (NIDA, 2017) with high co-occurring rates of IPV. The negative consequences are devastating to families and society. This team has developed a digital, interactive platform, RITch®CBT for the convenience of participants' within their own home & with out of session practice exercises. We propose to conduct a Phase I and II Study: UG3 (Phase I) and UH3 (Phase II) in collaboration with the FDA regarding ongoing feedback and regulatory processes. In Phase I, we propose a feasibility study, a randomized controlled trial to test the efficacy of RITch®CBT (n=20) among SUD-IPV diverse male clients entering addiction treatment comparing it to face to face 1:1 CBT (TAU, n=20). If efficacious, a Phase II (UH3, n=80) trial will be conducted to test the effectiveness of RITch®CBT among SUD-IPV compared to TAU (n=80) in reducing addiction and IPV.

DETAILED DESCRIPTION:
We propose to conduct a feasibility study across years 1-2 in collaboration with FDA's clinical data validation requirements to test the efficacy related endpoints of RITch®CBT by conducting a randomized trial. A total of 40 ethnically diverse male participants entering a substance abuse treatment facility, who meet current DSM-V criteria for substance dependence and have histories of IPV will be randomized to either "self-guided" 1:1 digital RITch®CBT Therapy (n=20) or 1:1 Standard CBT Therapy (n=20, non-digitized, 1:1 talk CBT). Each 60-minute session will occur 1x/week across 12 weeks of treatment.

* Primary outcomes will measure self-reported cravings via the AUC/DUC, number of days abstinent from substance use and number total days abstinent from aggression, both measured by the Timeline Follow-Back method, with confirmation via breath samples, urine toxicology screens, and verified by collateral reports.
* Primary Outcomes will be assessed at baseline, weekly through treatment, post-treatment, and at follow-ups 3, 6, and 9 months.
* Secondary outcome measures will be impulsivity and distress tolerance as measured by the Barratt Impulsiveness Scale (BIS) and Response to Conflict Scale (RTC), respectively.
* Tertiary outcomes will be Q-submissions, FDA feedback on regulatory pathways and IDE approval/confirmation of IDE required filings across the protocol.

ELIGIBILITY:
Inclusion Criteria:

Participants between the ages of 18-65 will be 40 men entering outpatient treatment who

(1) meet current DSM-V criteria substance dependence (and use alcohol and/or stimulants within the 30 days prior to the screening session); (2) report verbal aggression, conflict/aggression in a current intimate relationship (e.g., yelling, screaming, pushing, slapping) within 30 days prior to screening; and (3) can read English at a 6th grade level.

Exclusion Criteria:

Participants will be excluded if they: 1) Are currently in withdrawal from substance and in need of detoxification (such individuals may be re-evaluated following detoxification); 2) Have cognitive impairment (a mini mental state score <25); 3) Have psychomotor epilepsy (e.g. impulsivity or rage related symptoms secondary to a seizure disorder, as this medical diagnosis is likely to be a confound in the proposed study); 4) Have major medical complications such as a head injury/trauma, or HIV dementia that may also be a confound in the study interventions; 5) Are currently receiving either substance abuse or IPV treatment elsewhere; 6.) Have a lifetime history of any psychotic or bipolar disorder; or 7) Are currently suicidal or homicidal or 8) severe violence (punching, chocking, use of weapons).

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Substance Use Cravings | 84 days of treatment
  Self-reported cravings across 84 days as measured by the AUC/DUC

SECONDARY OUTCOMES:
Substance Use | 84 days
  Self report substance use across 84 days as measured by the Timeline Follow Back and verified by objective indicators of substance use (breathalyzer and urine toxicology screens)

CONTACTS AND LOCATIONS:
Overall Officials: James Filingeri, Study Chair — University of Rochester
Locations (1):
- Strong Recovery - Part Of Strong Memorial Hospital, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The proposed research may result in new technologies and methodologies to treat SUD and IPV. Since this study is a Phase I and II trial, and if results show that RITch®CBT is more effective than TAU in reducing Addiction and IPV, the data are intended to prepare this investigative team for a larger trial through dissemination across multiple sites. The data may also be applicable and useful to the community, the approaches and key results. Should there be requests for the raw datasets, these will be considered and we will be careful to review with our IRB and RRH CD clinic to ensure there is no possibility of violating the rights of any participants.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3-6 months after the study ends
Access Criteria: Caroline_Easton@URMC.Rochester.Edu
URL: http://www.rit.edu/favtech/contact-us

REFERENCES:
- [Background] Easton CJ, Crane CA, Mandel D. A Randomized Controlled Trial Assessing the Efficacy of Cognitive Behavioral Therapy for Substance-Dependent Domestic Violence Offenders: An Integrated Substance Abuse-Domestic Violence Treatment Approach (SADV). J Marital Fam Ther. 2018 Jul;44(3):483-498. doi: 10.1111/jmft.12260. Epub 2017 Nov 6. PMID 29108096